CLINICAL TRIAL: NCT00074243
Title: A Phase I Trial Of CC-8490 For The Treatment Of Patients With Recurrent/Refractory High-Grade Gliomas
Brief Title: CC-8490 in Treating Patients With Recurrent or Refractory High-Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000343702; NCI-04-C-0035; NCT00071864 (obsolete NCT alias)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2006-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult glioblastoma; adult mixed glioma; adult brain stem glioma; recurrent adult brain tumor; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Glioma; Brain Neoplasms; Gliosarcoma | interventions — CC-8490

INTERVENTIONS:
Drug: CC-8490

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as CC-8490, work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of CC-8490 in treating patients who have recurrent or refractory high-grade gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of CC-8490 in patients with recurrent or refractory high-grade gliomas.
* Determine, preliminarily, the toxic effects of this drug in these patients.
* Determine the pharmacokinetics of this drug in these patients.

Secondary

* Determine, preliminarily, the potential anti-glioma activity of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral CC-8490 once daily on days 1 and 3-28 (course 1 only). Beginning with course 2 and for all subsequent courses, patients receive oral CC-8490 once daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of CC-8490 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, a total of 10 patients are treated at that dose.

Patients are followed within 2 weeks.

PROJECTED ACCRUAL: A total of 34 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed supratentorial malignant glioma, including any of the following:

  * Glioblastoma multiforme
  * Gliosarcoma
  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Anaplastic mixed oligoastrocytoma
  * Malignant glioma/astrocytoma not otherwise specified OR
* Clinical and radiographic diagnosis of progressive low-grade glioma
* Radiographically diagnosed infiltrating brain stem gliomas not amenable to biopsy allowed
* Recurrent or progressive disease as determined by 1 of the following:

  * CT scan or MRI within the past 21 days
  * Biopsy within the past 12 weeks
* Failed prior radiotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* More than 8 weeks

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 8 g/dL (transfusion allowed)

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 2 times upper limit of normal
* No significant active hepatic disease that would preclude study participation

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No significant active renal disease that would preclude study participation

Cardiovascular

* No significant active cardiac disease that would preclude study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No significant active psychiatric disease that would preclude study participation
* No other condition or laboratory abnormality that would preclude study participation
* Able to swallow capsules whole

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 2 weeks since prior interferon
* No concurrent immunotherapy

Chemotherapy

* At least 2 weeks since prior vincristine
* At least 3 weeks since prior procarbazine
* At least 4 weeks since prior temozolomide or carboplatin
* At least 6 weeks since prior nitrosoureas
* No other concurrent anticancer chemotherapy

Endocrine therapy

* At least 2 weeks since prior tamoxifen
* Concurrent steroids allowed provided dose has been stable for at least 5 days prior to study enrollment

Radiotherapy

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 2 weeks since prior resection of a recurrent or progressive tumor

Other

* At least 2 weeks since other prior non-cytotoxic therapy
* At least 4 weeks since other prior cytotoxic therapies
* More than 28 days since prior experimental study drugs
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Fine, MD, Principal Investigator — NCI - Neuro-Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States